CLINICAL TRIAL: NCT04711148
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study of Orelabrutinib in Patients With Relapsing-Remitting Multiple Sclerosis to Evaluate Efficacy, Safety, Tolerability, Pharmacokinetics, and Biological Activity
Brief Title: A Phase 2 Study of Orelabrutinib in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-CL-00112
Record Dates: First submitted 2021-01-08; First posted 2021-01-15 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — orelabrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): The Core Part：Participants receive placebo
  The OLE Part：Participants who have completed the Week 24 visit in the Core Part for continued treatment and collect additional long-term safety and efficacy data receive the low dose of orelabrutinib or any other dose as suggested from the Core part of the study.
  Interventions: Other: placebo; Drug: orelabrutinib
- orelabrutinib(low dose) (Experimental): The Core Part：Participants receive low dose orelabrutinib
  The OLE Part：Participants who have completed the Week 24 visit in the Core Part for continued treatment and collect additional long-term safety and efficacy data receive the low dose of orelabrutinib or any other dose as suggested from the Core part of the study.
  Interventions: Drug: orelabrutinib
- orelabrutinib(medium dose) (Experimental): The Core Part ：Participants receive medium dose orelabrutinib
  The OLE Part：Participants who have completed the Week 24 visit in the Core Part for continued treatment and collect additional long-term safety and efficacy data receive the low dose of orelabrutinib or any other dose as suggested from the Core part of the study.
  Interventions: Drug: orelabrutinib
- orelabrutinib (high dose) (Experimental): The Core Part：Participants receive high dose orelabrutinib
  The OLE Part：Participants who have completed the Week 24 visit in the Core Part for continued treatment and collect additional long-term safety and efficacy data receive the low dose of orelabrutinib or any other dose as suggested from the Core part of the study.
  Interventions: Drug: orelabrutinib

INTERVENTIONS:
Other: placebo — placebo
  Arms: placebo
Drug: orelabrutinib — Orelabrutinib is a white, round, uncoated tablet

SUMMARY:
This is a randomized, double-Blind, placebo-controlled Phase 2 Study of Orelabrutinib in Patients with Relapsing-Remitting Multiple Sclerosis.

DETAILED DESCRIPTION:
The study contains 2 parts: Core Part and an Open-label Extension (OLE) Part.

The Core Part is a randomized, double-blind, placebo-controlled, phase 2 study. Patients with RRMS will be randomly assigned to 1 of 4 treatment groups. placebo, orelabrutinib (low dose), orelabrutinib (medium dose) and orelabrutinib (high dose) at a 1:1:1:1 ratio.

The OLE part is an open-label, single treatment arm study to enroll patients who have completed the Week 24 visit in the Core Part for continued treatment and collect additional long-term safety and efficacy data.All patients will receive the low dose of orelabrutinib or any other dose as suggested from the Core part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 to 55 years of age at the time of signing the informed consent.
2. Are diagnosed with Relapsing Remitting Multiple Sclerosis (RRMS).
3. Are neurologically stable for ≥ 30 days prior to both Screening and Baseline.
4. One or more documented relapses within the 2 years before Screening
5. Have an EDSS score of 0 to 5.5 at Screening and Baseline (Day 1)
6. Women of childbearing potential must use effective method of contraception
7. Signed and dated informed consent
8. Patient currently participating in the Core Part who has completed the end of treatment visit and will be benefit from continued treatment per investigator's assessment. (OLE Part only)

Exclusion Criteria:

1. Diagnosed with progressive MS.
2. Disease duration > 10 years in participants with an EDSS ≤ 2.0 at Screening and Baseline (Day 1).
3. Immunologic disorder other than MS.
4. History or current diagnosis of other neurological disorders that may mimic MS.
5. History or current diagnosis of progressive multifocal leukoencephalopathy (PML).
6. History of myocardial infarction or cerebrovascular event within 6 months prior to Screening,
7. A history of attempted suicide within 6 months prior to Screening or a positive response to items 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening.
8. An episode of major depression within the last 6 months prior to Screening (clinically stable minor depression is not exclusionary).
9. History of cancer, except adequately treated basal cell or squamous cell carcinoma of the skin
10. Breastfeeding/lactating or pregnant women
11. Participants are excluded from participation in the study if taken prohibited medications/treatments.
12. Participation in any investigational drug study within 6 months or 5 half-lives of the investigational drug, whichever is longest, prior to Screening.
13. Permanent discontinuation from the Core Part due to AE/ SAE or abnormal abnormalities or conditions leading to permanent study drug discontinuation. (OLE Part only)
14. Patient who has new abnormality appeared in the Core Part. (OLE Part only)
15. Any significant change in the subject's medical history that would preclude administration of the study drug. (OLE Part only)
16. Clinically significant laboratory abnormalities from the most recently available test in the Core Part that would preclude administration of the study drug. (OLE Part only)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The cumulative number of new GdE T1 MRI brain lesions | up to 120 weeks
  To evaluate the efficacy of orelabrutinib on the cumulative number of new gadolinium-enhancing (GdE) T1 magnetic resonance (MRI) brain lesions versus placebo over 12 weeks of treatment.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability ] | up to 120 weeks
  To evaluate the safety and tolerability of orelabrutinib compared to placebo in the Core Part
ARR[efficacy] | up to 120 weeks
  Annualized relapse rate in the OLE Part

OTHER OUTCOMES:
Peak concentration (Cmax) | up to 120 weeks
  Dose Escalation Peak concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (5):
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - University of South Florida, Tampa, Florida
  - Consultants in Neurology LTD, Northbrook, Illinois
  - Neurology Associates, P.C., Lincoln, Nebraska
  - Premier Neurology, P.C., Greer, South Carolina
- China (13):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - The 1st Affiliated Hospital of Shanxi Medical University, Taiyuan, Shan'xi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Air Force Military Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Poland (7):
  - NZOZ Wielospecjalistyczna Poradnia Lekarska "Synapsis", Katowice
  - Prywatna Praktyka Lekarska, Katowice
  - Resmedica NZOZ Kielce, Kielce
  - MCD Medical, Krakow
  - Neuromed, Lublin
  - Nzoz "Neuro-Kard", Poznan
  - Wielospecjalistyczne Centrum Medyczne Ibismed, Zabrze
- Ukraine (17):
  - CE I.I.Mechnykov Dnipropetrovsk RC Hosp of Dnipropetrovsk RC Dept of Neurology, Dnipro
  - Medical Center of Dnipro State Medical University, Dnipro State Medical University, Dnipro
  - SI USSRI of Medical and Social Problems of Disabilities of MOHU, Dnipro
  - CNE Regional Clinical Hospital of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Institute of Neurology, Psychiatry and Narcology of NAMSU, Kharkiv
  - SI Institute of Neurology, Psychiatry and Narcology of NAMSU, Kharkiv
  - CIH Kharkiv City General Practice, Kharkiv
  - Medical Center of Limited Liability Company Medbud-Clinic, Kyiv
  - CNE of Lviv Reg Council Lviv Reg Clin Hospital Dept of Neurology D.Halytskyi Lviv NMU, Lviv
  - CNE City Clinical Hospital #5 of Lviv, Lviv
  - CNE Odesa Regional Clinical Hospital of Odesa Regional Council, Odesa
  - Medical Center of Limited Liability Company Health Clinic, Medical Clinical Research Center, Vinnytsia
  - Medical Center of Limited Liability Company Medical Center Saliutem, Vinnytsia
  - Municipal Non-profit Enterprise "City Hospital No.6" of Zaporizhzya City Council, Zaporizhzhia
  - CNE Zaporizhzhia RCH of ZRC Dept of Neurology #1, Zaporizhzhia
  - CNE Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhia
  - Medical Center of Limited Liability Company INET-09, Zaporizhzhya